CLINICAL TRIAL: NCT05454280
Title: A Randomized Controlled Trial of Post-Discharge Risk-Based Management in Patients Undergoing High-Risk Elective Major Cancer Operations (PRS II)
Brief Title: Post-Discharge Risk-Based Management in Patients Undergoing High-Risk Elective Major Cancer Operations (PRS II)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-1013; SURG-210 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Surgery; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Eligible adult patients with probable or histologically/cytologically confirmed, primary or recurrent, malignant neoplasms (any stage) scheduled to undergo elective major cancer surgery at FCCC who meet eligibility criteria will be stratified by procedure type and randomized to the Intervention Arm or Control Arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm: Standard Perioperative Management (Active Comparator): Patients in the Control Arm will receive standard post-discharge surveillance (i.e., usual care).
  Interventions: Procedure: Standard post-discharge surveillance
- Intervention Arm: Intensified Post-Discharge Surveillance (Experimental): Patients in the Intervention and Control Arms will be monitored
  * Through PDD 30 for postoperative deaths and complications (as defined by ACS NSQIP) and/or adverse events (as defined by CTCAE)
  * Through the end of the index hospitalization for ICU admission, postoperative LOS, return to operating room, and discharge to home.
  * Through PDD 90 for hospital readmission, QOL, and receipt of anti-neoplastic therapy
  Interventions: Procedure: Intensified post-discharge surveillance

INTERVENTIONS:
Procedure: Intensified post-discharge surveillance — * TCC Nurse Televisit at post-discharge day 1 and 7
  * Televisit with APP/Resident/Fellow between post-discharge day 3-5
  * Referral for home health nursing evaluation upon discharge
  Arms: Intervention Arm: Intensified Post-Discharge Surveillance
Procedure: Standard post-discharge surveillance — Patients in the Control Arm will receive standard post-discharge surveillance, as deemed appropriate/necessary by the surgeons caring for them at the time of hospital discharge.
  Arms: Control Arm: Standard Perioperative Management

SUMMARY:
This is a randomized trial of intensified post-discharge surveillance (Intervention Arm) versus standard post-discharge surveillance (Control Arm).

DETAILED DESCRIPTION:
Eligible adult patients with probable or histologically/cytologically confirmed, primary or recurrent, malignant neoplasms (any stage) scheduled to undergo elective major cancer surgery at FCCC who meet eligibility criteria will be stratified by procedure type and randomized to the Intervention Arm or Control Arm.

• Prior to discharge, patients who meet eligibility criteria at Second Registration will be confirmed for study eligibility and randomized. Patients in the Control Arm will receive standard post-discharge surveillance, as deemed appropriate/necessary by the surgeons caring for them at the time of hospital discharge.

Patients in the Intervention and Control Arms will be monitored

* Through PDD 30 for postoperative deaths and complications (as defined by ACS NSQIP) and/or adverse events (as defined by CTCAE)
* Through the end of the index hospitalization for ICU admission, postoperative LOS, return to operating room, and discharge to home.
* Through PDD 90 for hospital readmission, QOL, and receipt of anti-neoplastic therapy

ELIGIBILITY:
First Registration Inclusion Criteria:

* Age > 18 years at diagnosis
* ECOG performance status 0, 1, or 2, defined as

Grade ECOG 0 Fully active, able to carry on all pre-disease performance without restriction

1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours

   * Patients must have probable (i.e., clinically suspicious) or histologically/cytologically confirmed, primary or recurrent, malignant neoplasm, malignant neuroendocrine tumor, or carcinoma in situ (any stage).

Patients undergoing major operations to resect or treat known or suspected malignancies of the head and neck, chest, abdomen, genitourinary tract, or extremities are eligible. Patients undergoing biopsies, outpatient procedures, superficial resections of cutaneous malignancies, or purely palliative operations are not eligible.

These procedures are commonly performed in patients with malignant neoplasms, malignant neuroendocrine tumors, or carcinomas in situ, and are commonly "tracked" by hospitals and cancer centers participating in the ACS NSQIP Procedure Targeted option because they are often associated with higher rates of postoperative morbidity and mortality (compared to other, less complex cancer procedures).

* Patient must be scheduled for elective major cancer surgery (as listed in 4.1.4) at FCCC < 30 days after First Registration.

Elective surgery is defined as:

* Patient is scheduled to be brought from their home (or normal living environment) to FCCC on the day of the index surgery (or day prior as scheduled admission) AND
* Surgery is not scheduled as urgent or emergent

  * Ability to understand and willingness to sign a written informed consent and HIPAA consent document
  * Geographical accessibility and willingness to return to FCCC for all preoperative and postoperative study assessments.

First Registration Exclusion Criteria:

* Any condition that might interfere with the subject's participation in the study, compliance with study requirements, or in the evaluation of the study results.

Second Registration Inclusion Criteria:

A patient will be eligible for continued inclusion in this study only if ALL of the following criteria apply at the time of Second Registration (one to two days prior to anticipated discharge). No exceptions or waivers will be granted for patients who do not meet the eligibility criteria.

* Post

  * Elective (curative or palliative) major cancer surgery (as listed in 4.1.4 above) at the time of the index surgery (patient may have undergone more than one of these procedures) OR
  * Elective surgical procedure(s) listed as an option (i.e., CPT code) in the Surgical Risk Calculator webpage (patient may have undergone more than one of these procedures)

For the purposes of this study, the procedure that was performed with the highest estimated risk of DSC (as predicted by the Surgical Risk Calculator) will be denoted at the time of Second Registration as the "index procedure" performed during the "index surgery".

* Elective surgery < 30 days after First Registration.

Second Registration Exclusion Criteria:

* Status post elective surgical procedure(s) not listed as options in the Surgical Risk Calculator webpage. This includes patients whose scheduled procedure was suspended due to unexpected findings, such as carcinomatosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
30-day rate of readmission/visit to emergency department/death | 30 days
  The primary objective of this trial is to determine if intensified post-discharge surveillance leads to a 7% absolute risk reduction/35% relative risk reduction in the composite endpoint of 30-day rate of readmission/visit to emergency department/death compared to standard post discharge management in patients undergoing elective, high risk cancer operations.

SECONDARY OUTCOMES:
30-day rate of death | 30 days
  Secondary objectives of the study are to determine whether intensified post-discharge surveillance leads to a reduction in 30-day rate of death
30-day rate of hospital readmission after index surgery | 30 days
  Secondary objectives of the study are to determine whether intensified post-discharge surveillance leads to a reduction in 30-day rate of hospital readmission after index surgery
60-day rate of hospital readmission after index surgery | 60 days
  Secondary objectives of the study are to determine whether intensified post-discharge surveillance leads to a reduction in 60-day rate of hospital readmission after index surgery
90-day rate of hospital readmission after index surgery | 90 days
  Secondary objectives of the study are to determine whether intensified post-discharge surveillance leads to a reduction in 90-day rate of hospital readmission after index surgery
30-day rate of unplanned Emergency Department visits | 30 days
  Secondary objectives of the study are to determine whether intensified post-discharge surveillance leads to a reduction in 30-day rate of unplanned Emergency Department visits

CONTACTS AND LOCATIONS:
Overall Officials: Jason Castellanos, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No